CLINICAL TRIAL: NCT01252953
Title: REVEAL: Randomized EValuation of the Effects of Anacetrapib Through Lipid-modification. A Large-scale, Randomized Placebo-controlled Trial of the Clinical Effects of Anacetrapib Among People With Established Vascular Disease
Brief Title: REVEAL: Randomized EValuation of the Effects of Anacetrapib Through Lipid-modification
Acronym: REVEAL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTSUREVEAL1; 48678192 (Registry Identifier: ISRCTN); 2010-023467-18 (EudraCT Number)
Record Dates: First submitted 2010-11-24; First posted 2010-12-03 (Estimated); Results first posted 2018-05-04 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: vascular disease; lipids; cholesteryl ester transfer protein (CETP) inhibition; anacetrapib
MeSH Terms: conditions — Atherosclerosis; Vascular Diseases; Inhibition, Psychological | interventions — anacetrapib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anacetrapib (Experimental)
  Interventions: Drug: Anacetrapib
- Placebo anacetrapib (Placebo Comparator)
  Interventions: Drug: Placebo anacetrapib

INTERVENTIONS:
Drug: Anacetrapib — tablet, 100mg daily
  Arms: Anacetrapib
Drug: Placebo anacetrapib — tablet, 1 tablet daily
  Arms: Placebo anacetrapib

SUMMARY:
The Randomized EValuation of the Effects of Anacetrapib Through Lipid-modification (REVEAL) trial aims to determine whether lipid modification with anacetrapib 100mg daily reduces the risk of coronary death, myocardial infarction (MI) or coronary revascularization (collectively known as major coronary events) in patients with circulatory problems who have their Low-density Lipoprotein (LDL) cholesterol level treated with a statin.

DETAILED DESCRIPTION:
Sub-study: Does anacetrapib as a CETP inhibitor lead to mobilization of stem cells and enhance myocardial function via neoangiogenesis and tissue regeneration?

Following the main on-treatment part of the study, there was a further period of at least 2 years during which participants were followed-up by telephone, off treatment.

All participants stopped study treatment prior to February 2017 (results for the main-trial have been reported) and direct participant follow-up was completed in April 2019.

In the UK we will continue to collect information on health outcomes via central data registries and NHS sources for many years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged at least 50 at the time of initial invitation, and at least one of the following inclusion criteria must be satisfied:

  * History of MI; or
  * Cerebrovascular atherosclerotic disease (i.e. history of presumed ischaemic stroke or carotid revascularization); or
  * Peripheral arterial disease (i.e. history of non-coronary revascularization, including aortic aneurysm repair or graft); or
  * Diabetes mellitus with other evidence of symptomatic coronary heart disease (i.e. treatment or hospitalization for angina, or a history of coronary revascularization or acute coronary syndrome).

Exclusion Criteria:

* None of the following must be satisfied:

  * Acute MI, acute coronary syndrome or stroke within 4 weeks prior to Screening Visit or during Run-in (but such individuals may be entered later, if appropriate);
  * Planned coronary revascularization procedure within the next 6 months (such individuals may be entered later, if appropriate);
  * Definite history of chronic liver disease, or abnormal liver function (i.e. alanine transaminase (ALT) >2x the upper limit of normal (ULN)). Note: Individuals with a history of acute hepatitis are eligible provided this ALT limit is not exceeded;
  * Severe renal insufficiency (i.e. creatinine >200 µmol/L [2.3 mg/dL], dialysis or functioning renal transplant);
  * Evidence of active inflammatory muscle disease (e.g. dermatomyositis, polymyositis), or creatine kinase (CK) >3x ULN;
  * Previous significant adverse reaction to a statin or anacetrapib;
  * Current treatment with any of the following lipid-lowering treatments:

    (i) a regimen considered to produce substantially greater LDL cholesterol reduction than atorvastatin 80 mg daily for individuals in non-Asian countries or 20 mg daily for those in North East Asia; or (ii) fibric acid derivative ("fibrate", including gemfibrozil); or (iii) niacin (nicotinic acid) at doses above 100 mg daily
  * Concurrent treatment with a medication that is contraindicated with anacetrapib or atorvastatin:

    (i) any potent CYP3A4 inhibitor, such as:
    1. macrolide antibiotics (erythromycin, clarithromycin, telithromycin);
    2. systemic imidazole or triazole antifungals (e.g. itraconazole, posaconazole);
    3. protease inhibitors (e.g. atazanavir);
    4. nefazodone

       (ii) ciclosporin

       (iii) daptomycin

       (iv) systemic use of fusidic acid

       Note: Individuals who are taking such drugs temporarily may be re-screened when they discontinue them, if considered appropriate;
  * Known to be poorly compliant with clinic visits or prescribed medication;
  * Medical history that might limit the individual's ability to take trial treatments for the duration of the study (e.g. severe respiratory disease; history of cancer or evidence of spread within last 5 years, other than non-melanoma skin cancer; or recent history of alcohol or substance misuse);
  * Women of child-bearing potential (unless using adequate contraception);
  * Current participation in a clinical trial with an unlicensed drug or device.

Individuals will also be excluded at the Screening visit if it is considered unlikely that they will achieve total cholesterol <3.5 mmol/L (135 mg/dL) on the highest atorvastatin dose available in their region (atorvastatin 80 mg daily in non-Asian countries or 20 mg daily in North East Asia).

In addition, individuals will be excluded at the Randomization visit if any of the following are true:

* Total cholesterol above 4 mmol/L [155 mg/dL]
* Non-compliant with run-in treatment (<90% scheduled run-in medication taken)
* Individual is no longer willing to be randomized into the 4-5 year trial
* The individual's doctor is of the view that their patient should not be randomized.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30449 (Actual)
Dates: Start 2011-06; Primary Completion 2017-01-31 (Actual); Study Completion 2037-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Landray, Principal Investigator — University of Oxford; Louise Bowman, Principal Investigator — University of Oxford
Locations (1):
- CTSU, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Proposals for substudies must be approved by the Steering Committee. Procedures for accessing the data for this study are available on: https://www.ndph.ox.ac.uk/data-access.
Supporting Information: Study Protocol, SAP
Access Criteria: See URL
URL: https://www.ndph.ox.ac.uk/data-access

REFERENCES:
- [Background] REVEAL Collaborative Group; Bowman L, Chen F, Sammons E, Hopewell JC, Wallendszus K, Stevens W, Valdes- Marquez E, Wiviott S, Cannon CP, Braunwald E, Collins R, Landray MJ. Randomized Evaluation of the Effects of Anacetrapib through Lipid-modification (REVEAL)-A large-scale, randomized, placebo-controlled trial of the clinical effects of anacetrapib among people with established vascular disease: Trial design, recruitment, and baseline characteristics. Am Heart J. 2017 May;187:182-190. doi: 10.1016/j.ahj.2017.02.021. Epub 2017 Feb 21. PMID 28454801
- [Result] HPS3/TIMI55-REVEAL Collaborative Group; Bowman L, Hopewell JC, Chen F, Wallendszus K, Stevens W, Collins R, Wiviott SD, Cannon CP, Braunwald E, Sammons E, Landray MJ. Effects of Anacetrapib in Patients with Atherosclerotic Vascular Disease. N Engl J Med. 2017 Sep 28;377(13):1217-1227. doi: 10.1056/NEJMoa1706444. Epub 2017 Aug 28. PMID 28847206
- [Result] Hopewell JC, Ibrahim M, Hill M, Shaw PM, Braunwald E, Blaustein RO, Bowman L, Landray MJ, Sabatine MS, Collins R; HPS3/TIMI55-REVEAL Collaborative Group. Impact of ADCY9 Genotype on Response to Anacetrapib. Circulation. 2019 Sep 10;140(11):891-898. doi: 10.1161/CIRCULATIONAHA.119.041546. Epub 2019 Jul 23. PMID 31331193
- [Result] HPS3/TIMI55-REVEAL Collaborative Group; Writing Committee; Sammons E, Hopewell JC, Chen F, Stevens W, Wallendszus K, Valdes-Marquez E, Dayanandan R, Knott C, Murphy K, Wincott E, Baxter A, Goodenough R, Lay M, Hill M, Macdonnell S, Fabbri G, Lucci D, Fajardo-Moser M, Brenner S, Hao D, Zhang H, Liu J, Wuhan B, Mosegaard S, Herrington W, Wanner C, Angermann C, Ertl G, Maggioni A, Barter P, Mihaylova B, Mitchel Y, Blaustein R, Goto S, Tobert J, DeLucca P, Chen Y, Chen Z, Gray A, Haynes R, Armitage J, Baigent C, Wiviott S, Cannon C, Braunwald E, Collins R, Bowman L, Landray M; REVEAL Collaborative Group. Long-term safety and efficacy of anacetrapib in patients with atherosclerotic vascular disease. Eur Heart J. 2022 Apr 6;43(14):1416-1424. doi: 10.1093/eurheartj/ehab863. PMID 34910136
- [Result] Lui JNM, Williams C, Keng MJ, Hopewell JC, Sammons E, Chen F, Gray A, Bowman L, Landray SMJ, Mihaylova B; REVEAL Collaborative Group. Impact of New Cardiovascular Events on Quality of Life and Hospital Costs in People With Cardiovascular Disease in the United Kingdom and United States. J Am Heart Assoc. 2023 Oct 3;12(19):e030766. doi: 10.1161/JAHA.123.030766. Epub 2023 Sep 26. PMID 37750555
- [Derived] Landmesser U, von Eckardstein A, Kastelein J, Deanfield J, Luscher TF. Increasing high-density lipoprotein cholesterol by cholesteryl ester transfer protein-inhibition: a rocky road and lessons learned? The early demise of the dal-HEART programme. Eur Heart J. 2012 Jul;33(14):1712-5. doi: 10.1093/eurheartj/ehs182. Epub 2012 Jun 13. No abstract available. PMID 22696435
- [Derived] Krauss RM, Wojnooski K, Orr J, Geaney JC, Pinto CA, Liu Y, Wagner JA, Luk JM, Johnson-Levonas AO, Anderson MS, Dansky HM. Changes in lipoprotein subfraction concentration and composition in healthy individuals treated with the CETP inhibitor anacetrapib. J Lipid Res. 2012 Mar;53(3):540-547. doi: 10.1194/jlr.M018010. Epub 2011 Dec 17. PMID 22180633
- See also: REVEAL trial website — https://www.revealtrial.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized between August 2011 and October 2013. Follow-up continued until 31st January 2017.
Pre-assignment Details: Successfully screened participants were entered into a run-in period. Attendees were discouraged from continuing to randomization if it was thought unlikely they would be able to continue attending follow-up visits for at least 4-5years. During run-in participants were issued atorvastatin (1 tablet/day) and placebo anacetrapib (1 tablet/day).
Groups:
- Anacetrapib: Anacetrapib: 100mg tablet daily
- Placebo Anacetrapib: Placebo anacetrapib: 1 tablet daily
Period: Overall Study
Arm/Group | Anacetrapib | Placebo Anacetrapib
Started | 15225 | 15224
Completed | 15187 | 15186
Not Completed | 38 | 38
Not completed — Withdrawal by Subject | 16 | 17
Not completed — Lost to Follow-up | 22 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anacetrapib | Placebo Anacetrapib | Total
Number analyzed (Participants) | 15225 | 15224 | 30449
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6634 | 6643 | 13277
  >=65 years | 8591 | 8581 | 17172
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (8) | 67 (8) | 67 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2456 | 2459 | 4915
  Male | 12769 | 12765 | 25534
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 121 | 114 | 235
  Not Hispanic or Latino | 2560 | 2522 | 5082
  Unknown or Not Reported | 12544 | 12588 | 25132
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 160 | 168 | 328
  Race: Chinese | 4323 | 4323 | 8646
  Race: Other North East Asian | 5 | 6 | 11
  Race: South Asian | 95 | 97 | 192
  Race: South East Asian | 11 | 11 | 22
  Race: White | 10561 | 10558 | 21119
  Race: Other | 47 | 49 | 96
  Race: Mixed | 21 | 12 | 33
  Race: Unknown | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4204 | 4177 | 8381
  Norway | 426 | 418 | 844
  Sweden | 427 | 434 | 861
  Denmark | 918 | 932 | 1850
  Finland | 307 | 306 | 613
  Germany | 755 | 774 | 1529
  Italy | 826 | 834 | 1660
  United States | 2687 | 2643 | 5330
  Canada | 361 | 391 | 752
  China | 4314 | 4315 | 8629
Previous disease [Count of Participants; unit: Participants] — The participants could have more than one of these conditions.
  Participants
    Coronary heart disease | 13325 | 13354 | 26679
    Cerebrovascular disease | 3385 | 3396 | 6781
    Peripheral-artery disease | 1229 | 1206 | 2435
    Diabetes | 5654 | 5666 | 11320
    Heart failure | 902 | 869 | 1771
Region [Count of Participants; unit: Participants]
  Europe | 7863 | 7875 | 15738
  North America | 3048 | 3034 | 6082
  China | 4314 | 4315 | 8629
Systolic Blood Pressure, Categorical [Count of Participants; unit: Participants]
  <125 mmHg | 5678 | 5760 | 11438
  ≥125 to <140 mmHg | 4819 | 4740 | 9559
  ≥140 mmHg | 4728 | 4724 | 9452
Systolic Blood Pressure, Continuous [Mean (Standard Deviation); unit: mmHg] | 131.3 (18.5) | 131.1 (18.5) | 131.2 (18.5)
Diastolic Blood Pressure, Categorical [Count of Participants; unit: Participants]
  < 75 mmHg | 5656 | 5790 | 11446
  ≥ 75 to < 85 mmHg | 5408 | 5277 | 10685
  ≥ 85 mmHg | 4161 | 4157 | 8318
Diastolic Blood Pressure, Continuous [Mean (Standard Deviation); unit: mmHg] | 78.1 (10.9) | 78.0 (11.0) | 78.1 (11.0)
Body Mass Index, Categorical [Count of Participants; unit: Participants] — The body mass index is the weight in kilograms divided by the square of the height in meters.
  Participants
    <25 kg/m^2 | 3447 | 3361 | 6808
    ≥25 to < 30 kg/m^2 | 6949 | 6995 | 13944
    ≥ 30 kg/m^2 | 4829 | 4868 | 9697
Body Mass Index, Continuous [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (5.0) | 28.6 (5.1) | 28.6 (5.1)
LDL Cholesterol, Categorical [Count of Participants; unit: Participants]
  < 54 mg/dl | 5023 | 5077 | 10100
  ≥ 54 to < 66 mg/dl | 4643 | 4705 | 9348
  ≥ 66 mg/dl | 5559 | 5442 | 11001
LDL Cholesterol, Continuous [Mean (Standard Deviation); unit: mg/dl] | 61 (15) | 61 (15) | 61 (15)
Non-HDL Cholesterol, Categorical [Count of Participants; unit: Participants]
  < 85 mg/dl | 5642 | 5701 | 11343
  ≥ 85 to <101 mg/dl | 4896 | 4853 | 9749
  ≥ 101 mg/dl | 4687 | 4670 | 9357
Non-HDL Cholesterol, Continuous [Mean (Standard Deviation); unit: mg/dl] | 92 (19) | 92 (19) | 92 (19)
HDL Cholesterol, Categorical [Count of Participants; unit: Participants]
  < 35 mg/dl | 4583 | 4590 | 9173
  ≥ 35 to < 43 mg/dl | 5438 | 5269 | 10707
  ≥ 43 mg/dl | 5204 | 5365 | 10569
HDL Cholesterol, Continuous [Mean (Standard Deviation); unit: mg/dl] | 40 (10) | 40 (10) | 40 (10)
Glomerular Filtration Rate, Categorical [Count of Participants; unit: Participants] — The estimated glomerular filtration rate was calculated with the use of the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation as per Levey AS, Stevens LA, Schmid CH, et al. A new equation to estimate glomerular filtration rate.
  Ann Intern Med 2009; 150(9): 604-12.
  Participants
    < 60 ml/min/1.73m^2 | 1655 | 1698 | 3353
    ≥ 60 ml/min/1.73m^2 | 13570 | 13526 | 27096
Glomerular Filtration Rate, Continuous [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 83 (17) | 83 (17) | 83 (17)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Coronary Event
Description: Primary assessment involves an intention-to-treat comparison among all randomized participants of the effects of allocation to anacetrapib versus placebo on major coronary events (defined as the occurrence of coronary death, myocardial infarction or coronary revascularization procedure) during the scheduled treatment period.
  Data reported is for the first major coronary event.
Time Frame: Randomized treatment phase during median follow-up period of 4.1years
Measure: Count of Participants; unit: Participants
Arm/Group | Anacetrapib | Placebo Anacetrapib
Number analyzed (Participants) | 15225 | 15224
Participants | 1640 | 1803
Statistical Analysis 1: Comparison: Anacetrapib vs Placebo Anacetrapib; Test type: Other — Time to first event; p = 0.004, Log Rank; Rate Ratio = 0.91, 95% CI 2-sided [0.85 to 0.97]

2. Secondary Outcome: Number of Participants With Major Atherosclerotic Event
Description: Major atherosclerotic events (defined as coronary death, myocardial infarction or presumed ischaemic stroke; the key secondary outcome).
  Secondary assessments involve intention-to-treat comparisons among all randomized participants of the effects of allocation to anacetrapib versus placebo during the scheduled treatment period.
Time Frame: Randomized treatment phase during median follow-up period of 4.1years
Measure: Count of Participants; unit: Participants
Groups:
- Anacetrapib: Anacetrapib: 100mg daily
Arm/Group | Anacetrapib | Placebo Anacetrapib
Number analyzed (Participants) | 15225 | 15224
Participants | 1383 | 1483
Statistical Analysis 1: Comparison: Anacetrapib vs Placebo Anacetrapib; Test type: Other — Time to first event; p = 0.052, Log Rank; Rate Ratio = 0.93, 95% CI 2-sided [0.86 to 1]

3. Secondary Outcome: Number of Participants With Presumed Ischaemic Stroke
Description: Presumed ischaemic stroke (i.e. not known to be haemorrhagic).
  Secondary assessments involve intention-to-treat comparisons among all randomized participants of the effects of allocation to anacetrapib versus placebo during the scheduled treatment period.
Time Frame: Randomized treatment phase during median follow-up period of 4.1years
Measure: Count of Participants; unit: Participants
Arm/Group | Anacetrapib | Placebo Anacetrapib
Number analyzed (Participants) | 15225 | 15224
Participants | 485 | 489
Statistical Analysis 1: Comparison: Anacetrapib vs Placebo Anacetrapib; Test type: Other — Time to first event; In accordance with the data analysis plan, if the outcome of a major atherosclerotic event did not reach significance, there was no hypothesis testing for presumed ischemic stroke, so no P value is given; Rate Ratio = 0.99, 95% CI 2-sided [0.87 to 1.12]

4. Secondary Outcome: Number of Participants With Major Vascular Event
Description: Major vascular events (defined as coronary death, myocardial infarction, coronary revascularization or presumed ischaemic stroke).
  Secondary assessments involve intention-to-treat comparisons among all randomized participants of the effects of allocation to anacetrapib versus placebo during the scheduled treatment period
Time Frame: Randomized treatment phase during median follow-up period of 4.1years
Measure: Count of Participants; unit: Participants
Arm/Group | Anacetrapib | Placebo Anacetrapib
Number analyzed (Participants) | 15225 | 15224
Participants | 2068 | 2214
Statistical Analysis 1: Comparison: Anacetrapib vs Placebo Anacetrapib; Test type: Other — Time to first event; p = 0.02, Log Rank; Rate Ratio = 0.93, 95% CI 2-sided [0.88 to 0.99]

ADVERSE EVENTS:
Time Frame: Randomized treatment phase during median follow-up period of 4.1years
Description: All participants were assessed for adverse events at 6-monthly intervals at which relevant information was recorded on the electronic case report form. In accordance with the protocol, Serious Adverse Events were recorded for all participants (30,449 subjects) and non-serious Adverse Events (presented in the 'Other Adverse Events' section) were recorded in North America only (6,082 subjects).
Arm/Group | Anacetrapib | Placebo Anacetrapib
All-Cause Mortality (participants affected / at risk) | 1122/15225 | 1155/15224
Serious Adverse Events (participants affected / at risk) | 8898/15225 | 8912/15224
Other Adverse Events (participants affected / at risk) | 2493/3048 | 2503/3034
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anacetrapib (N=15225) | Placebo Anacetrapib (N=15224)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 188 (219) | 182 (210)
Cardiac disorders (Cardiac disorders) | 2568 (4120) | 2766 (4280)
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 9 (9) | 4 (4)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 114 (121) | 91 (99)
Endocrine disorders (Endocrine disorders) | 50 (50) | 49 (51)
Eye disorders (Eye disorders) | 204 (235) | 232 (264)
Gastrointestinal disorders (Gastrointestinal disorders) | 813 (1012) | 788 (976)
General disorders & administration site conditions (General disorders) | 691 (781) | 736 (838)
Hepatobiliary disorders (Hepatobiliary disorders) | 217 (251) | 238 (268)
Immune system disorders (Immune system disorders) | 12 (12) | 29 (29)
Infections and infestations (Infections and infestations) | 1559 (2097) | 1537 (2152)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 753 (889) | 777 (918)
Investigations (Investigations) | 1105 (1421) | 1135 (1419)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 642 (774) | 687 (820)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 438 (508) | 432 (501)
Neoplasms benign, malignant and unspecified (incl cycts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1323 (1810) | 1295 (1770)
Nervous system disorders (Nervous system disorders) | 1399 (1789) | 1455 (1822)
Psychiatric disorders (Psychiatric disorders) | 104 (117) | 111 (124)
Renal and urinary disorders (Renal and urinary disorders) | 415 (516) | 398 (470)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 49 (53) | 56 (59)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 606 (791) | 605 (813)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 84 (93) | 97 (109)
Social circumstances (Social circumstances) | 501 (769) | 516 (778)
Surgical and medical procedures (Surgical and medical procedures) | 3409 (5051) | 3478 (5241)
Vascular disorders (Vascular disorders) | 346 (399) | 352 (393)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anacetrapib (N=3048) | Placebo Anacetrapib (N=3034)
Cardiac disorders (Cardiac disorders) | 169 | 208
Eye disorders (Eye disorders) | 227 | 230
Gastrointestinal disorders (Gastrointestinal disorders) | 596 | 557
General disorders and administration site conditions (General disorders) | 321 | 338
Infections and infestations (Infections and infestations) | 974 | 943
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 480 | 516
Investigations (Investigations) | 327 | 307
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 405 | 393
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1125 | 1105
Nervous system disorders (Nervous system disorders) | 625 | 623
Psychiatric disorders (Psychiatric disorders) | 155 | 139
Renal and urinary disorders (Renal and urinary disorders) | 160 | 171
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 463 | 412
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 203 | 211
Surgical and medical procedures (Surgical and medical procedures) | 211 | 202
Vascular disorders (Vascular disorders) | 185 | 189

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-01-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT01252953/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT01252953/SAP_001.pdf